CLINICAL TRIAL: NCT03342209
Title: Determination of Half-life of the Carboxyhemoglobin Level and Utility of High Flow Nasal Cannula in Carbon Monoxide Toxicity in the Emergency Department
Brief Title: Utility of High Flow Nasal Cannula in CO Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ibrahim Ulas Ozturan, Principle Investigator, MD, Kocaeli University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIA 2016/286
Record Dates: First submitted 2017-10-28; First posted 2017-11-14 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2017-11

CONDITIONS: Carbon Monoxide Poisoning; Environmental Exposure
Keywords: carbon monoxide toxicity; high flow nasal cannula; emergency department
MeSH Terms: conditions — Carbon Monoxide Poisoning; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HFNC therapy (Experimental): Fisher&Paykel AIRVO™ 2 High Flow Nasal Cannula Therapy will be implemented to CO-poisoned patients. Oxygen flow rate will be started 60 L/min and be decreased as the patient has requested.
  Interventions: Device: Fisher&Paykel AIRVO™ 2 High Flow Nasal Cannula Therapy

INTERVENTIONS:
Device: Fisher&Paykel AIRVO™ 2 High Flow Nasal Cannula Therapy — A high flow nasal cannula will be implemented to the CO-poisoned patients. In the meantime, intravenous access and cardiac monitorization will have been establishing. When the high flow nasal cannula becomes ready, the first venous blood sample will be taken and the treatment will be started without any delay. The gas flow rate will be started at the rate of 30 liters per minute and will be increased to the max flow rate which patient can tolerate and FiO2 of 1.0. If the first COHb level is lesser than 10%, the patient will be excluded and will receive standard emergency care.
  The blood sample will be drawn from existing IV access every 10 minutes until the COHb levels become %50 or lesser of the initial level.
  Once the COHb level becomes 50% of initial measurement, following blood samples will be taken in every 30 minutes.

SUMMARY:
determination of the half-life of COHb in CO-poisoned patients with high flow nasal oxygen therapy in the ED.

DETAILED DESCRIPTION:
Carbon monoxide (CO) poisoning is common and potentially fatal environmental emergency which requires immediate attention. It is responsible for up to 40,000 emergency department (ED) visits and 5000 to 6000 deaths per year, making it one of the leading causes of poisoning death in the United States. The management options for CO poisoning are limited to high flow oxygen by face mask or hyperbaric oxygen treatment. While half-life of carboxyhemoglobin (COHb) in a patient treating with high flow oxygen via a nonbreathing face mask is 90 minutes, it becomes 30 minutes with hyperbaric oxygen treatment (HBO).

The hypothesis of this study is using high flow nasal oxygen therapy in the CO poisoning may be more effective and safer treatment method comparing to standard oxygen therapy in the ED. Also, it may be a safe promising alternative of hyperbaric oxygen therapy.

The aim of the study is to determine the half-life of COHb in CO-poisoned patients with high flow nasal oxygen therapy in the ED.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are admitted to the emergency department with CO poisoning with a CoHB level of >10%.
* The patients who accept to participate in the study.

Exclusion Criteria:

* The patients who are <18 years old.
* The patients who need mechanical ventilation
* The patients who are implemented oxygen more than 30 minutes before the ED admission
* The patients who will be transferred to the hyperbaric oxygen center before the CoHB levels are decreased to the half.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Half life of COHb | between 20 and 120 minutes
  Half life of COHb levels (%) under the high flow nasal oxygen therapy. Elimination rate of COHb will be determined in every 10 minutes according to venous blood gas COHb level.

SECONDARY OUTCOMES:
Adverse Events | between 0 and 120 minutes
  Mucosal dryness, epistaxis and burn in the nasal cavity will be evaluated as a adverse events of high flow nasal cannula.
Device Comfort | Between 0 and 120 minutes
  Patient comfort will be assessed according to verbal numeric rating scale by asking to patient to say a number between 0 to 10 with 0 being "high flow nasal cannula can not be tolerated" and 10 being " the most comfortable breath ever".
Flow Rate Tolerability | Between 0 and 120 minutes
  Flow rate tolerability will be assessed according to patient request to change in flow rate.
Flow Temperature Tolerability | Between 0 and 120 minutes.
  Flow temperature tolerability will be assessed according to patient request to change in flow rate.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yaka, Assoc. Prof., Study Chair — Kocaeli University; İbrahim U Özturan, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University Medical Faculty, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided